CLINICAL TRIAL: NCT03162302
Title: Free-Breathing Liver Fat and Iron Quantification Using 3D Stack-of-Radial MRI
Brief Title: Liver Fat and Iron Quantification MRI
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Holden H. Wu, PhD, Associate Professor-in-Residence, University of California, Los Angeles
Other Study IDs: 17-000276
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Liver Diseases
Keywords: MRI; magnetic resonance imaging; fat quantification; iron quantification
MeSH Terms: conditions — Liver Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Healthy volunteers will undergo 60 minute non-contrast enhanced Magnetic Resonance Imaging (MRI) of the abdomen using novel imaging sequences.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Clinical Patients: Patients in whom an MRI is indicated for their disease condition will undergo the clinical scan, followed by up to 30 minutes non-contrast enhanced Magnetic Resonance Imaging (MRI) of the abdomen using novel imaging sequences. Clinical patients may also elect to undergo a research only scan of approximately one hour.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Magnetic resonance imaging (MRI) is a non-invasive imaging technique that uses a magnetic field and radio waves to create detailed images of the organs and tissues within the body.
  Other Names: MR

SUMMARY:
The objective of this study is to develop and evaluate novel magnetic resonance imaging (MRI) protocols for studying the structure and function of the human body using 1.5 Tesla and 3.0 Tesla MRI scanners with or without the use of an MRI contrast agent.

DETAILED DESCRIPTION:
This study will include on-going technical development work for the non-invasive diagnosis of liver fat or iron accumulation and other abnormalities. MRI is a non-invasive imaging technique with no known side effects. The study will utilize imaging equipment that is used routinely in numerous hospitals and clinics around the world.

The project seeks to address optimization of the imaging methodology at 1.5 Tesla and 3.0 Tesla in the liver and abdomen in order to improve clinical evaluation and care of future patients. Non contrast MRI studies will be performed in normal healthy subjects. In addition, the study will include subjects with confirmed disease or who have suspicion for disease, and are undergoing contrast or non-contrast MR imaging as part of their standard of care. Up to sixty-five (65) male or female subjects eighteen years of age and older will be studied in total (number includes healthy subjects and non-healthy subjects).

Currently, clinical MRI exams are of adequate spatial and temporal resolution, sufficient quantitative accuracy, and acceptable exam duration, but improvements in each of these areas would benefit the care of future patients. For example, improvements in spatial and temporal resolution may confer greater conspicuity of disease and shortening the exam duration can be expected to improve patient acceptance and minimize motion artifacts. The study explores innovative ideas about ways to improve MRI exams to have impact in all three of these areas.

Current MRI techniques for fat and iron quantification in the liver and abdomen are challenged by respiratory and organ motion. As a result, imaging parameters (coverage, resolution, etc) and TE (echo time) selection for fat/iron quantification are compromised to accommodate a short breath-held 2D or 3D scan, which can still be affected by motion artifacts and even unachievable for patients with limited breath-holding capability. Therefore, the study aims to achieve robust free-breathing fat/iron quantification in the liver and abdomen using innovative MRI techniques and algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers:

   * Healthy subjects 18 years or older
2. Clinical Patients:

   * Patients who are 18 years or older and who are scheduled for a routine clinically indicated MRI exam at University of California Los Angeles

Exclusion Criteria:

1. Healthy Volunteers:

   * Age less than 18 years
   * Subject with the following devices/implants/conditions will be excluded:

     1. cardiac pacemakers
     2. defibrillators
     3. cochlear implants
     4. intraocular metallic foreign bodies
     5. intracranial aneurysm clips
     6. claustrophobia
   * Subjects will be excluded if they have a history of severe renal disease (Creatinine level >2.5 mg/dl or Glomerular Filtration Rate <15 ml/minute/1.73m2 ) or allergy to MRI contrast agents ("dyes"). Healthy volunteers will not be studied with these agents.
   * Pregnant subjects will not be enrolled. Although there is no data to suggest that MRI is harmful to the fetus, this study is limited to non-pregnant subjects.
2. Clinical Patients:

   * Age less than 18 years
   * Subject with the following devices/implants/conditions will be excluded:

     1. cardiac pacemakers
     2. defibrillators
     3. cochlear implants
     4. intraocular metallic foreign bodies
     5. intracranial aneurysm clips
     6. claustrophobia
   * Subjects will be excluded if they have a history of severe renal disease (Creatinine level >2.5 mg/dl or Glomerular Filtration Rate <15 ml/minute/1.73m2 ) or allergy to MRI contrast agents ("dyes").
   * Pregnant subjects will not be enrolled. Although there is no data to suggest that MRI is harmful to the fetus, this application is limited to non-pregnant subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll healthy volunteers over age 18 and clinical patients who are scheduled to undergo a clinically indicated MRI of the abdomen or who are willing to undergo a separate research scan.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Proton Density Fat Fraction (0 to 100%) in the liver of each subject | 2 years
  MRI based measurement of liver fat content using proton density fat fraction
Transverse Magnetization Relaxation Rate R2* (1/sec) in the liver of each subject | 2 years
  MRI based measurement of R2* is associated with underlying liver iron content

CONTACTS AND LOCATIONS:
Overall Officials: Holden H Wu, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No